CLINICAL TRIAL: NCT04482959
Title: Intraoperative Carbetocin to Decrease Blood Loss During Hysteroscopic Myomectomy: a Randomized Controlled Trial
Brief Title: Intraoperative Carbetocin to Decrease Blood Loss During Hysteroscopic Myomectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Taman, lecturer, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MS.20.07.1178
Record Dates: First submitted 2020-07-19; First posted 2020-07-23 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Myoma;Uterus
MeSH Terms: conditions — Myofibroma | interventions — carbetocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial (RCT).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization will be simple and balanced (1:1) and will be carried out by a nurse through sealed, unlabeled, opaque envelopes containing computer-generated random numbers. The participants, caregivers and investigators will be blinded to group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbetocin group (Experimental): This group will contain 20 patients having single type 0 or I submucous uterine myomas according to International Federation of Gynecology and Obstetrics classification system with a largest diameter ≤ 4 cm and myometrial free margin of at least 10 mm.After induction of general anesthesia, immediately before the operation, participants will receive either 1 ml of carbetocin (100 mcg/ml) IV over 1 minute.
  Interventions: Drug: Carbetocin
- • Control group (Placebo Comparator): This group will contain 20 patients having single type 0 or I submucous uterine myomas according to International Federation of Gynecology and Obstetrics classification system with a largest diameter ≤ 4 cm and myometrial free margin of at least 10 mm.After induction of general anesthesia, immediately before the operation, participants will receive either 1 ml of sodium chloride 0.9% IV over 1 minute.
  Interventions: Drug: Sodium chloride 0.9%

INTERVENTIONS:
Drug: Carbetocin — (1-deamino-1-monocarba-(0-2-methyltyrosine)-oxytocin) is a long-acting synthetic agonist analogue of the human oxytocin
  Arms: Carbetocin group
Drug: Sodium chloride 0.9% — Physiological solution will be used as placebo
  Arms: • Control group

SUMMARY:
Submucous myomas represent one of the main indications of operative hysteroscopy. Since 1976 when Neuwirth and Amin reported the first five cases of excision of submucous myomas , several techniques have been developed in order to render hysteroscopic myomectomy a safe and effective procedure .

Hysteroscopic myomectomy is currently considered the "gold standard" minimally invasive approach for the treatment of symptomatic submucous myomas . Patients undergoing hysteroscopic myomectomy are liable to significant blood loss, and hemodynamic and hematological disturbances. Excessive bleeding during hysteroscopic myomectomy remains a major challenge for the endoscopic gynecological surgeons. Many interventions were introduced to reduce the risk of bleeding during myomectomy. These include the use of utero-tonics such as oxytocin, or the use of anti-fibrinolytics such as tranexamic acid . The potential advantage of oxytocin infusion during hysteroscopic myomectomy is that it can maintains uterine contractility throughout the procedure, and thus, reduce blood loss .

Carbetocin (1-deamino-1-monocarba-(0-2-methyltyrosine)-oxytocin) is a long-acting synthetic agonist analogue of the human oxytocin. When injected to a woman, it induces uterine contractions . Although many interventions have been described to reduce the intraoperative blood loss during hysteroscopic myomectomy, there is a need for a well-designed randomized controlled trials to identify the most efficient interventions, with reasonable safety profiles, to help the perform a safe and curative surgery.

DETAILED DESCRIPTION:
All patients will have preoperative evaluation by gynecologists and anesthetists, with history taking and pelvic examination. A TVS scan will be done to determine the number, size and location of the myomas, and evaluate the myometrial free margin (the minimum thickness between the outer edge of the myoma and inner edge of the uterine serosa), which was found to be ideally ≥ 10 mm (11). Prior office diagnostic hysteroscopy will be performed for evaluation of the number, location and grade of the submucous myomas, and assessment of the endocervical canal and uterine cavity and the position of the tubal ostia in order to aid orientation. Preoperative full blood count, serum creatinine, fasting blood glucose, liver enzymes, coagulation profile ( INR), and viral markers will be done for all the patients. Monopolar resectoscopic myomectomies will be scheduled in the proliferative phase of menstrual cycle by a single experienced operator.

After induction of general anesthesia, immediately before the operation, participants will receive either 1 ml of carbetocin (100 mcg/ml) IV over 1 minute (study group) or 1 ml of sodium chloride 0.9% IV over 1 minute (control group). The procedure will be done using the available standard setup and the distending solution used will be 1.5% glycine. A drape with a fluid-collection pouch (Lingeman 3 in 1 Procedure Drape, Lingeman Medical Products, Inc., Indianapolis, IN) placed beneath the woman's buttocks will be used to collect outflow fluid escaping between the cervix and sheath to prevent spillage of irrigating fluid onto the floor. Fluid inflow and outflow will be monitored every 3-5 minutes. The outflow fluid will be measured to the nearest milliliter. The inflow and outflow volumes of the distension solution will be carefully monitored continuously during the procedure by nurses not involved in the study under the current monitoring protocol at the operating theater. The procedure would be terminated if the fluid imbalance reached 1 L.

After completing the procedure, the surgeon completed a record sheet for rating of bleeding amount and the quality of operative view. Postoperative full blood count will be done for all patients 24 hours after the procedures. Preoperative and postoperative hemoglobin and hematocrit, the need for blood transfusion, the duration of operation, any operative complications and medication adverse effects will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic women aged 18-45 years diagnosed by transvaginal sonography (TVS) to have single type 0 or I submucous uterine myomas according to FIGO classification system with a largest diameter ≤ 4 cm and myometrial free margin of at least 10 mm.

Exclusion Criteria:

* • Age < 18 or > 45 years.

  * Uterine septum or structural uterine abnormality (including multiple uterine fibroids and/or multiple submucous myomas)
  * Present or history of cervical or uterine malignancies.
  * Active pelvic infection.
  * Chronic medical diseases (cardiopulmonary, thromboembolic, hepatic, or renal diseases).
  * Bleeding disorders.
  * Patients receiving anticoagulant therapy.
  * Patients receiving gonadotropin-releasing hormone (GnRH) analogues.
  * History of adverse reaction contraindications for Carbetocin.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding amount | Time Frame: Start with the first resectoscope myoma cut till withdrawal of hysteroscope through the cervix at the end of the procedure
  Minimal Bleeding is insufficient to interfere with the operation or with the clarity of vision Moderate Bleeding that obscure the visual field and resolves only with continuous and constant irrigation of the distention media Excessive Bleeding that necessitate intervention other than continuous and constant irrigation of the distention media (e.g. controlled only by increasing the pressure to tamponade the bleeding from myoma bed)
• Change in haemoglobin and hematocrit | Haemoglobin and hematocrit values 24 hours before myomectomy and 24 hour after myomectomy
  • Change in haemoglobin and hematocrit as surrogate measures of haemostatic effect

SECONDARY OUTCOMES:
• Operative time | Start with insertion of hysteroscope through the cervix ends with withdrawal of hysteroscopy through the cervix at the end of the procedure
  It evaluate the complication that could affect the technique
• Fluid deficit | start with insertion of hysteroscope through the cervix ends with withdrawal of hysteroscopy through the cervix at the end pf the procedure
  Calculation the fluid deficit between in flow volume and outflow volume.
• The quality of operative view | start with the first resectoscope myoma cut till the completion of myoma resection
  Poor When it is not possible to visualize the entire uterine cavity and the cornual areas nor adequate visualization of the myoma during more than half of the procedure despite continuous and constant irrigation of the distention media Fair When it is not possible to visualize the entire uterine cavity and the cornual areas nor adequate visualization of the myoma during less than half of the procedure despite continuous and constant irrigation of the distention media Good When it is possible to assess the entire uterine cavity to include the cornual areas from the level of isthmus satisfactorily throughout the entire procedure with adequate visualization of the myoma.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed E Taman, MD, Principal Investigator — Faculty of Medicine - Mansoura University
Locations (1):
- Faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neuwirth RS, Amin HK. Excision of submucus fibroids with hysteroscopic control. Am J Obstet Gynecol. 1976 Sep 1;126(1):95-9. doi: 10.1016/0002-9378(76)90471-3. PMID 961753
- [Result] Di Spiezio Sardo A, Mazzon I, Bramante S, Bettocchi S, Bifulco G, Guida M, Nappi C. Hysteroscopic myomectomy: a comprehensive review of surgical techniques. Hum Reprod Update. 2008 Mar-Apr;14(2):101-19. doi: 10.1093/humupd/dmm041. Epub 2007 Dec 6. PMID 18063608
- [Result] Deutsch A, Sasaki KJ, Cholkeri-Singh A. Resectoscopic Surgery for Polyps and Myomas: A Review of the Literature. J Minim Invasive Gynecol. 2017 Nov-Dec;24(7):1104-1110. doi: 10.1016/j.jmig.2017.08.645. Epub 2017 Aug 24. PMID 28843536
- [Result] Malm M, Madsen I, Kjellstrom J. Development and stability of a heat-stable formulation of carbetocin for the prevention of postpartum haemorrhage for use in low and middle-income countries. J Pept Sci. 2018 Jun;24(6):e3082. doi: 10.1002/psc.3082. Epub 2018 Apr 27. PMID 29700898
- [Result] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435